CLINICAL TRIAL: NCT03338530
Title: Efficacy of a Comprehensive School-based Intervention for High-functioning Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canisius College (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-13#142RENEWAL-Ammend
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Psychosocial treatment; School intervention; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The efficacy of the comprehensive school-based intervention (CSBI) was evaluated in a cluster randomized trial (pretest-posttest control group design). School buildings were randomly assigned to receive the CSBI or their typical educational programming. The CSBI was examined for its effect on the social performance/competence, ASD symptoms, and academic skills of children with HFASD compared to children with HFASD that did not receive the intervention. School staff delivered the multi-component intervention during the school year and research staff monitored intervention implementation (fidelity).
Who Masked: Outcomes Assessor
Masking Description: Child testing and behavioral observations were completed by evaluators blinded to treatment condition; evaluators consisted of advanced graduate students with training in the specific outcome measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive School-Based Intervention (Experimental): Children with HFASD assigned to the CSBI received social skills groups, computer instruction in emotion recognition, therapeutic activities, and a behavioral reinforcement system (individual daily note) during the school year and their parents participated in monthly parent training. School staff received training prior to the school year and demonstrated fidelity with the protocol. Fidelity was also monitored during the school year by research assistants.
  Interventions: Behavioral: Comprehensive School-Based Intervention
- Business-As-Usual (BAU) Control (No Intervention): Children with HFASD in the BAU schools received their typical special education programming as legally-mandated. The programming received by each was carefully monitored per the following: 1) Each student's IEP was reviewed to document the legally mandated services received; 2) For those receiving counseling or speech-language services, the related-service provider completed a survey indicating specific treatment targets and the protocol for service provision; 3) Parents completed a monthly survey of any external therapeutic programming their child may have received; and 4) Fidelity measures designed for the intervention group (with sequencing requirements removed) were completed for the control condition during two 60-minute classroom observations per week by research assistants.

INTERVENTIONS:
Behavioral: Comprehensive School-Based Intervention — School staff administered the 5 components during the school year. Social Skills Groups were conducted 2-3x/wk. for a total of 60-90 min./wk.; each group contained 3-6 students with social impairments. The Individual Daily Note was administered across the school day to reinforce new skills and reduce problem symptoms. Students' performance on targets was linked to home rewards. Mind Reading computer instruction targeting emotion recognition skills was conducted 3x/wk. for a total of 60 min./wk. Therapeutic Activities were conducted 2x/wk. for a total of 40-60 min./wk.; these cooperative activities were designed to practice targeted skills. Parent Training was conducted 1x/month for 60-90 min./session in order to increase home-school communication and integrate the CSBI across settings.
  Arms: Comprehensive School-Based Intervention

SUMMARY:
This study was a 4-year efficacy trial (cluster randomized trial) of a comprehensive school-based intervention (CSBI) for high-functioning elementary students with autism spectrum disorder (HFASD). The sample included children, in grades 1-5 with HFASD enrolled in public schools. School buildings were randomly assigned to either receive the CSBI or serve as the control comparison (business-as-usual [BAU]). School staff in the CSBI schools administered social skills groups (60-90 minutes per week), facial-emotion recognition computer instruction (60 minutes per week), therapeutic activities (40-60 minutes per week), a behavioral reinforcement system (across the school day), and parent training (60-90 minutes per month) during the school year. Children with HFASD in the BAU schools received their typical educational program. Implementation fidelity was assessed by research assistants throughout the school year in the CSBI schools using standardized fidelity monitoring sheets. The fidelity monitoring sheets were also completed by research assistants during observations in the BAU schools in order to identify the possible presence of any of the treatment elements in the control (BAU) schools. Outcome measures were completed for both groups at baseline (6 weeks into the school year prior to the initiation of the intervention) and at the end of the school year following completion of the intervention. Primary outcome measures included a test of emotion recognition and parent-teacher ratings of ASD symptoms and secondary measures included parent-teacher ratings of social/social-communication skills, a test of academic achievement skills, and a direct behavioral measure of social interaction skills (child testing and behavioral observations were completed by evaluators blinded to treatment condition; parent-teacher raters were not blinded to treatment condition). For the primary measures/analyses, it was hypothesized that students with HFASD who complete the CSBI will demonstrate significantly greater emotion-recognition skills and receive significantly lower parent-teacher ratings of ASD symptoms compared to controls. For the secondary measures/analyses, it was hypothesized that students with HFASD who complete the CSBI will receive significantly higher parent-teacher ratings of social/social-communication skills, demonstrate significantly higher academic skills, and exhibit significantly higher rates of social interactions with peers compared to controls.

DETAILED DESCRIPTION:
The efficacy of the comprehensive school-based intervention (CSBI) was evaluated in a cluster randomized trial (pretest-posttest control group design). A total of 96 students in grades 1-5 with HFASD from 32 public elementary schools were initially targeted for enrollment over the 4-year study period. Once students were screened and determined to meet eligibility criteria, individual schools (clusters) were randomly assigned to either the treatment condition (CSBI) or control condition (business-as-usual [BAU]). A block randomization design with stratification by school economic level was used to insure approximate balance among the treatment groups. Recruitment was conducted during the 4-8 months prior to the upcoming school year. School staff from the treatment schools completed a manualized 5-day training during the summer preceding the treatment year and demonstrated fidelity with the protocol (competence). Pretesting was completed 6 weeks into the school year (prior to the initiation of the intervention) and posttesting at the end of the school year following completion of the intervention. Children with HFASD in the CSBI schools received the CSBI intervention implemented by school staff during the school year and children with HFASD in the BAU schools received their typical special education programming. Implementation accuracy (fidelity) was assessed by research assistants throughout the school year in the CSBI schools using standardized fidelity monitoring sheets. The fidelity monitoring sheets were also completed by research assistants during observations in the BAU schools in order to identify the possible presence of any of the treatment elements in the BAU schools.

Treatment (CSBI) group protocol. The following is a description of the 5 treatment components (SSGs, IDN, MR, TAs, and PT) and fidelity protocol for the CSBI.

Social skills groups (SSGs). SSGs were conducted 2-3x/wk. for a total of 60-90 min./wk. by a designated member of the school team. Groups contained 3-6 students with social impairments. Each manualized SSG began with a review of rules and was then conducted according to the framework of Skillstreaming (Goldstein et al., 1997). Skillstreaming is a structured program for teaching interpersonal skills to children with social deficits using teaching, modeling, role-playing, performance feedback, and transfer of learning (McGinnis & Goldstein, 1997). In the CSBI, 26 social skills were taught in a progression from basic to more complex. While the SSG protocol required active participation of every child each session, each child was required to be the primary role-player at least twice per 3 sessions. Each session ended with a short review and discussion of how to use the skill in future classroom activities. To ensure repeated practice and ongoing feedback, and promote generalization, 1) each participant had >2 social targets on her/his IDN (see IDN section), 2) classroom teachers displayed a list of the social skills taught to date and the component steps of each social skill, and 3) parents were continually informed of target skills. Fidelity of implementation. SSG facilitators recorded the date, attendees, minutes of group instruction, and skill for each session on a tracking sheet and research assistants monitored fidelity at least 1x/wk. using a standardized fidelity sheet.

Individual daily note (IDN). The IDN was administered across the school day and was used to practice and reinforce newly learned skills, and reduce problem behaviors/ASD symptoms. It directed the student, school team, and parents to focus on specific skills/behaviors and performance criteria, and promoted communication between school and home. Each IDN consisted of 3-5 operationally-defined targets; to increase generalization >2 were skills taught in the CSBI. Initially, IDN targets were identified by teachers and operationally defined, and base rate data were collected for 3-5 days to determine criteria for IDN goals. Each student's school day was then divided into intervals based on his/her reinforcement needs. At the end of each interval, the student could earn 1 point for each IDN target and must have earned >75% of her/his daily points to receive a home reward (reinforcer). During each interval, the student received immediate verbal feedback and a tally was recorded on his/her IDN. At the end of each interval, the teacher provided feedback on the student's performance during that interval based on the targets and performance criteria. At the end of the day, the teacher informed the student of her/his overall performance (% earned), sent a copy of the IDN home, and retained a copy of the IDN. Fidelity of implementation. A copy of each child's IDN was kept by the classroom teacher and collected every 2 weeks. Adherence was assessed during at least two 60-min. observations each week using a standardized fidelity sheet.

Mind Reading (MR) computer instruction. MR was conducted 3x/wk. for a total of 60 min./wk. by a designated member of the school team. MR is an interactive software program designed to teach recognition of emotions in facial and vocal formats (Baron-Cohen et al., 2004). It features 412 emotions organized into 24 emotion groups and by 6 emotion levels. The program presents instruction and tasks in the Emotions Library, Learning Center, and Games Zone and reinforcing activities in the Rewards Zone. It also employs a token system to reinforce participants with access to the Rewards Zone using points earned for accurate completion of questions in MR. The CSBI included 100 MR emotions divided into 10 groups (10 emotions per group). Each week students were taught 1 group of emotions (repeated during the 3 lessons). After each emotion group was taught, students repeated the 10 emotion groups 2 more times for a total of 3 exposures to the 10 groups. Each session was manualized to ensure children met time parameters accessing areas of MR. School staff members monitored students to ensure they accessed program areas according to the protocol. Fidelity of implementation. Data on time using the software for each participant were collected by an internal chronometer in the software and research assistants monitored implementation accuracy at least once per week using a standardized fidelity sheet.

Therapeutic activities (TAs). TAs were conducted 2x/wk. for a total of 40-60 min./wk. by a designated member of the classroom team. TAs required >2 students and were conducted to practice and reinforce social skills and face-emotion recognition, and promote interest expansion. Each TA was written as a lesson plan that described the activity, its purpose, skill targeted, materials needed, deficit addressed, and procedures for conducting the activity. TAs were conducted with general and/or special education peers. At the outset, facilitators reviewed the activity rules and quickly discussed the activity. The facilitator also discussed with the target student how she/he can use the target and previously taught skills during the activity. During TAs, facilitators maintained proximity to the target students and provided frequent reinforcement when students exhibited target skills and corrective feedback when necessary. Each TA ended with a quick debriefing (1-3 min.) including how students used target skills during the TA and how they can use these skills during the school day/week. Fidelity of implementation. TA facilitators recorded the date, attendees, minutes of instruction, and skill targeted for each session on a tracking sheet. Research assistants monitored fidelity at least 3x/month using a standardized fidelity sheet.

Parent training (PT). PT was conducted 1x/month for 60-90 min./session during the school year by at least 1 member of the school team. This served to increase home-school communication and integrate the CSBI across settings. It also fostered active parent participation in the establishment of home reinforcers for school performance on treatment targets and increased parental understanding of the CSBI. PT content and instructional procedures were manualized to ensure delivery of consistent content. Facilitators delivered content using detailed lesson plans and PowerPoint slides or showed a video recording of the session(s) (which covered the same lesson plans and PowerPoints). Each session was structured as follows: 1) Brief updates on CSBI and PT agenda; 2) Lesson content (delivered live or via video); 3) Discussion of content and integration of content into daily routine; and 4) Review of session content and implementation procedures. Fidelity of implementation. PT facilitators recorded the date, attendees, duration of session, and topic covered for each session on a tracking sheet. Research assistants monitored fidelity at least 1x per 2 PT sessions using a standardized fidelity sheet.

Consultation support. Consultants provided support for classroom teams via weekly meetings. Consultants generally consisted of graduate students with advanced training in assessment and treatment of ASD/HFASD. Most were recruited from prior psychosocial treatment trials for children with HFASD conducted by our team and, as such they had extensive training and experience in administering the active components of the CSBI, and the fidelity, data collection, and data entry procedures. Fidelity of implementation. Consultants met with teams at least 1x/wk. and documented meetings on a log which included the school/team, date, time, topic(s), and outcome. The logs were reviewed monthly and child progress was reviewed at weekly consultant case review meetings with the study's clinical director.

Comparison (BAU) group protocol. Research indicates that students with HFASD do not receive adequate, intensive, or comprehensive school interventions (White, Scahill et al., 2007). This suggested that students randomly assigned to the control (BAU) condition would not receive services that remotely approximated the intensity or scope of the CSBI. Given randomization at the school level, contamination was unlikely however we monitored the roles of school staff and excluded any staff member (e.g., related-service provider) who provided services across buildings. The services received by the control children (programming and services mandated on their IEPs) were also monitored to ensure they were sufficiently different from the CSBI group. Four procedures were used. 1) Each student's IEP was reviewed to identify and document the legally mandated services she/he received. 2) For those receiving counseling (group or individual) or speech-language services, the related-service provider completed a survey indicating specific treatment targets and the protocol for service provision (techniques used, number of trials, etc.). 3) Parents completed a monthly survey of any external therapeutic or social-communicative programming their child may have received. 4) Fidelity measures designed for the intervention group (with sequencing requirements removed) were completed for the control condition during two 60-minute classroom observations per week by research assistants.

ELIGIBILITY:
Inclusion Criteria: (1) WISC-IV short form IQ>70 (and VCI or PRI>80); (2) CASL expressive or receptive language score >75; and (3) a score meeting ASD criteria on the ADI-R

Exclusion Criteria: Evidence of psychosis

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cambridge Mindreading Face-Voice Battery for Children (CAM-C) Scores at Follow-up | Baseline (immediately prior to treatment) and follow-up (immediately following treatment)
  Total score used to assess emotion recognition skills; scores range from 0 to 90, with higher scores indicating better emotion recognition accuracy/skills
Change from Baseline Social Responsiveness Scale, 2nd Edition, School Age Form (SRS-2) Scores at Follow-up | Baseline (immediately prior to treatment) and follow-up (immediately following treatment)
  SRS-2 total composite score normative mean = 50 and standard deviation = 10, with higher scores indicating more severe autism spectrum disorder symptoms/impairments

SECONDARY OUTCOMES:
Change from Baseline Adapted Skillstreaming Checklist (ASC) Scores at Follow-up | Baseline (immediately prior to treatment) and follow-up (immediately following treatment)
  Total ASC score used to assess social/social-communication skills; scores range from 38 to 190, with higher scores indicating greater use of social/social-communication skills
Change from Baseline Woodcock-Johnson III Tests of Achievement (WJ III ACH) Scores at Follow-up | Baseline (immediately prior to treatment) and follow-up (immediately following treatment)
  Standard scores (mean = 100 and standard deviation = 15) used from the Letter Word Identification, Calculation, Spelling, Passage Comprehension, and Writing Samples subtests, with higher scores indicating better academic skills
Change from Baseline Social Interaction Observation Scale (SIOS) Scores at Follow-up | Baseline (immediately prior to treatment) and follow-up (immediately following treatment)
  Total SIOS score used to measure the frequency of social interactions during social activities, with higher total scores indicating more social interactions

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Lopata, PsyD, Principal Investigator — Institute for Autism Reseach, Canisius College

IPD SHARING:
Plan to Share IPD: Undecided
We are evaluating the appropriate means to make the data available to other researchers (e.g., NDAR)

REFERENCES:
- [Background] Goldstein, A. P., McGinnis, E., Sprafkin, R. P., Gershaw, N. J., & Klein, P. (1997). Skillstreaming the adolescent: New strategies and perspectives for teaching prosocial skills, revised edition. Champaign, IL: Research Press.
- [Background] McGinnis, E., & Goldstein, A. P. (1997). Skillstreaming the elementary school child: New strategies and perspectives for teaching prosocial skills, revised edition. Champaign, Il: Research Press.
- [Background] Baron-Cohen, S., Golan, O., Wheelwright, S., & Hill, J. J. (2004). Mind reading: The intervention guide to emotions. London: Jessica Kingsley Limited (www.jkp.com).
- [Background] White SW, Scahill L, Klin A, Koenig K, Volkmar FR. Educational placements and service use patterns of individuals with autism spectrum disorders. J Autism Dev Disord. 2007 Sep;37(8):1403-12. doi: 10.1007/s10803-006-0281-0. Epub 2006 Nov 3. PMID 17082975
- [Background] Golan O, Baron-Cohen S. Systemizing empathy: teaching adults with Asperger syndrome or high-functioning autism to recognize complex emotions using interactive multimedia. Dev Psychopathol. 2006 Spring;18(2):591-617. doi: 10.1017/S0954579406060305. PMID 16600069
- [Background] Constantino, J. N., & Gruber, C. P. (2012). Social Responsiveness Scale, Second Edition (SRS-2). Torrance, CA: Western Psychological Services.
- [Background] Lopata C, Thomeer ML, Volker MA, Nida RE, Lee GK. Effectiveness of a manualized summer social treatment program for high-functioning children with autism spectrum disorders. J Autism Dev Disord. 2008 May;38(5):890-904. doi: 10.1007/s10803-007-0460-7. PMID 18058012
- [Background] Lopata C, Thomeer ML, Volker MA, Toomey JA, Nida RE, Lee GK, Smerbeck AM, Rodgers JD. RCT of a manualized social treatment for high-functioning autism spectrum disorders. J Autism Dev Disord. 2010 Nov;40(11):1297-310. doi: 10.1007/s10803-010-0989-8. PMID 20232240
- [Background] Woodcock, R. W., McGrew, K. S., & Mather, N. (2001). Woodcock-Johnson III Tests of Achievement. Itasca, IL: Riverside Publishing.
- [Background] Bauminger N. The facilitation of social-emotional understanding and social interaction in high-functioning children with autism: intervention outcomes. J Autism Dev Disord. 2002 Aug;32(4):283-98. doi: 10.1023/a:1016378718278. PMID 12199133
- [Background] Wechsler, D. (2003). Wechsler Intelligence Scale for Children (4th ed.). San Antonio, TX: The Psychological Corporation.
- [Background] Carrow-Woolfolk, E. (1999). Comprehensive Assessment of Spoken Language. Circle Pines, MN: American Guidance Services.
- [Background] Rutter, M., LeCouteur, A., & Lord, C. (2003). Autism Diagnostic Interview-Revised. Los Angeles: Western Psychological Services.
- [Derived] Lopata C, Thomeer ML, Rodgers JD, Donnelly JP, Lodi-Smith J. Longitudinal Follow-Up Study of Social Intervention Outcomes for Children on the Autism Spectrum. J Autism Dev Disord. 2025 Feb;55(2):393-407. doi: 10.1007/s10803-023-06221-1. Epub 2024 Feb 8. PMID 38326493
- [Derived] Lopata C, Thomeer ML, Rodgers JD, Donnelly JP, McDonald CA, Volker MA, Smith TH, Wang H. Cluster Randomized Trial of a School Intervention for Children with Autism Spectrum Disorder. J Clin Child Adolesc Psychol. 2019 Nov-Dec;48(6):922-933. doi: 10.1080/15374416.2018.1520121. Epub 2018 Oct 30. PMID 30376652